CLINICAL TRIAL: NCT02196103
Title: Management of Labor in Patients With Previous Cesarian Section and Premature Rupture of Membranes Who Desire TOLAC: Comparison Between the Use of Standard Expectant Management and the Double-balloon Catheter Device. A Prospective Randomized Study
Brief Title: Management of Labor in Patients With Previous Cesarian Section
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0019-14-HYMC
Record Dates: First submitted 2014-07-15; First posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Pregnancy; Previous Cesarian Section; Premature Rupture of Membranes (PROM)
Keywords: TOLAC; PROM; Previous Cesarian section; Mechanical cervical ripening
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Expectant management (Experimental)
  Interventions: Device: Double balloon cervical catheter

INTERVENTIONS:
Device: Double balloon cervical catheter

SUMMARY:
Induction of labor in women desiring TOLAC has long been a topic of controversy. The paucity of published data on mechanical cervical ripening in the setting of TOLAC and term PROM has led us to undertake the present clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed to be pregnant with PROM at >34 weeks. Rupture of membranes will be determine clinically and confirmed by positive Nitrazine test.
* Ruptured membranes have occurred in the last 24 hours prior to inclusion in the study.
* Found to have an unripe cervix in a speculum examination.
* Singleton pregnancy in a vertex presentation well applied to the cervix and absence of significant and regular uterine contractions (3-5/10 Min)
* Previous on cesarian section.
* Willingness to comply with the protocol for the duration of the study.
* Have signed an informed consent.

Exclusion Criteria: Patients having any of the following conditions:

* Any contraindication for the vaginal delivery (i.e. placenta previa, non vertex presentation).
* Regular uterine contractions (3-5/10 min).
* Diagnosis of rupture membranes was made over 24 hours prior the study inclusion.
* Evidence of chorio-amnionitis (T 37.6 celsious Degree with uterine tenderness and maternal or fetal tachycardia or purulent discharge or WBC>/=20,000)
* Suspected placental abruption or presence of a significant hemorrhage.
* Non-reassuring fetal status (as determined by fetal heart rate monitoring and/or bio-physical profile) necessitating immediate intervention.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
vaginal delivery rate | 48 hours
  20% higher vaginal delivery rate

SECONDARY OUTCOMES:
safety | 48 hours
  safety of the double balloon device in women with one previous cesarian section and PROM at >/=34 weeks by monitoring fetal heart rate, increased uterine hemorrhage, maternal hemodinamic changes, and uterine atony.

OTHER OUTCOMES:
satisfaction | 48 hours
  maternal experience and satisfaction with the method of delivery that was applied

CONTACTS AND LOCATIONS:
Overall Officials: Asnat Walfisch, MD, Principal Investigator — Hillel Yaffe Medical Center

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264